CLINICAL TRIAL: NCT01312207
Title: Macular Tractional Retinoschisis in Proliferative Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chung-May Yang, National Taiwan University Hospital
Other Study IDs: 201101020RC
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: tractional retinoschisis; traction retinal detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: To evaluate the clinical manifestations and surgical prognosis of macular tractional retinoschisis in proliferative diabetic retinopathy.

Design: Retrospective case series. Participants: Cases with macular tractional retinoschisis with or without combined traction detachment (TRD) in proliferative diabetic retinopathy confirmed by optical coherence tomography (OCT) at a single institution between January 2007 and August 2010.

Methods: Cases were divided into two groups. Group A had tractional retinoschisis only while Group B had TRD with retinoschisis of the elevated retina. Clinical data including OCT findings were recorded and analyzed.

Main Outcome Measures: Demographic data, clinical pictures, surgical results, and OCT findings will be compared between two the groups.

DETAILED DESCRIPTION:
Fibrovascular tissue induced macular elevation is an important cause of visual loss in proliferative diabetic retinopathy (PDR). There are two main types of macular elevations in PDR: traction retinal detachment (TRD) and tractional retinoschisis. These two conditions may coexist either in the form of retinoschisis within the detached retina or predominantly retinoschisis with a small subfoveal fluid pocket. Optical coherence tomography (OCT) studies have shown that in tractional retinoschisis, the inner retinal layer is normal reflective; outer layer is less reflective but not optically empty. Bridging columnar tissues are frequently observed between the inner and outer layers. Histopathological study by Faulborn et al showed adherence of posterior hyaloid membrane to the retina plus vitreous body shrinkage might induce retinal elevation with splitting of the outer plexiform layer, leading to retinoschisis. The bridging columnar tissues between inner and outer layers of the split retina mainly consisted of Muller cells. Although tractional retinoschisis with or without retinal detachment has been suggested as the most frequent pattern of tractional macular elevation in eyes with proliferative diabetic retinopathy1, and peripheral retinoschisis are frequently found during operation for complications of PDR, studies on clinical manifestations and post-operative visual prognosis of macular traction schisis are limited. Lincoff reported a relatively good prognosis in eyes with tractional retinoschisis after vitrectomy. No other large series specifically aimed at this entity can be found.

In this report, we will retrospectively study the clinical pictures of tractional retinoschisis on the macula. Morphological changes and functional outcomes after surgery will be discussed. Correlations between visual acuity and specific findings on color fundus pictures and OCT will be evaluated. We will also analyze different behaviors of schisis only and combined tractional retinal detachment with schisis.

ELIGIBILITY:
Inclusion Criteria:

tractional retinoschisis without TRD in PDR tractional retinoschisis with TRD in PDR

Exclusion Criteria:

active vitreous hemorrhage

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases with macular tractional retinoschisis with or without combined traction detachment (TRD) in proliferative diabetic retinopathy confirmed by optical coherence tomography
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-08 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
visual acuity change after surgery | before surgery and 3 months after surgery
  visual acuity (in logMAR ) before and after surgery

SECONDARY OUTCOMES:
Optical coherence tomography findings | before and after surgery
  schisis pattern and assocaiated macular changes after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chung-May Yang, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Imai M, Iijima H, Hanada N. Optical coherence tomography of tractional macular elevations in eyes with proliferative diabetic retinopathy. Am J Ophthalmol. 2001 Sep;132(3):458-61. doi: 10.1016/s0002-9394(01)01176-x. PMID 11530091
- [Background] Faulborn J, Ardjomand N. Tractional retinoschisis in proliferative diabetic retinopathy: a histopathological study. Graefes Arch Clin Exp Ophthalmol. 2000 Jan;238(1):40-4. doi: 10.1007/s004170050007. PMID 10664051